CLINICAL TRIAL: NCT04338854
Title: The Evaluation of The Effect of Routine Treatments Administrated in Pedodontics Clinics on Dental Anxiety in Children and Salivary Cortisol Levels
Brief Title: Dental Anxiety in Children and Salivary Cortisol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burçin Acar, Principal Investigator, Inonu University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-840
Record Dates: First submitted 2020-02-10; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Dental Anxiety
Keywords: dental anxiety; cortisol; procedure
MeSH Terms: interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Root canal treatment (Experimental): It's one of the restorative groups with LA (Local Anesthesia). An aerator and micromotor were used as cavity preparation in this group. Only conventional root canal treatment and extirpation were planned for the children included in the root canal treatment group in the measurement session.
  Interventions: Procedure: Restorative Treatment
- Pulpotomy treatment (Experimental): It's one of the restorative groups with LA (Local Anesthesia).An aerator and micromotor were used as cavity preparation in this group. it was noted that at least one of the approximal surfaces of the teeth had decay and iron sulfate (ViscoStat®, UltraDent, South Jordan, USA) was used as pulpotomy material
  Interventions: Procedure: Restorative Treatment
- two-surface restoration with Local Anesthesia (Experimental): It's one of the restorative groups with LA (Local Anesthesia).An aerator and micromotor were used as cavity preparation in this group. A Tofflemire matrix retainer and 0.05 mm thick matrix band (Hahnenkratt, Königsbach-Stein, Germany) were used in groups with a two-surface cavity.
  Interventions: Procedure: Restorative Treatment
- one surface restoration with Local Anesthesia (Experimental): It's one of the restorative groups with LA (Local Anesthesia).An aerator and micromotor were used as cavity preparation in this group.
  Interventions: Procedure: Restorative Treatment
- two-surface restoration without Local Anesthesia (Experimental): An aerator and micromotor were used as cavity preparation in this group. A Tofflemire matrix retainer and 0.05 mm thick matrix band (Hahnenkratt, Königsbach-Stein, Germany) were used in groups with a two-surface cavity.
  Interventions: Procedure: Restorative Treatment
- one surface restoration without Local Anesthesia (Experimental): An aerator and micromotor were used as cavity preparation in this group.
  Interventions: Procedure: Restorative Treatment
- fluoride application by disposable arch tray (Experimental): It's one of the protective groups.Only the micromotor was used for polishing purposes in the protective treatment groups. 2% NaF (Polimo® IMICRYL, Konya, Turkey) was preferred in groups who received fluoride application.
  Interventions: Procedure: Restorative Treatment
- fluoride application by cotton roll (Experimental): It's one of the protective groups. Only the micromotor was used for polishing purposes in the protective treatment groups 2% NaF (Polimo® IMICRYL, Konya, Turkey) was preferred in groups who received fluoride application.
  Interventions: Procedure: Restorative Treatment
- Fissure Sealant group (Experimental): It's one of the protective groups. Only the micromotor was used for polishing purposes in the protective treatment groups.
  Interventions: Procedure: Restorative Treatment

INTERVENTIONS:
Procedure: Restorative Treatment — 9 groups were formed as 6 restorative and 3 protective applications. The restorative treatment groups included procedures with- and without-local anesthesia (LA). Procedures with LA included the groups as root canal treatment, pulpotomy, two-surface restoration and one-surface restoration. Procedures without LA included the groups as two-surface restoration and one-surface restoration. The protective application groups included the groups as fluoride application (by disposable arch tray or by cotton roll) and fissure sealant.
  Other Names: Protective Application

SUMMARY:
Objective: This study aimed to assess whether pediatric dental anxiety is due to the day of dental appointment, to the dental chair, or to the dental treatment procedure during the course of the first dental treatment in children.

Study Design: Salivary cortisol samples were taken on three sequential days (pre-treatment, treatment and post-treatment days) and during the beginning and at ~15th minute of treatment, and at 15th minute post-treatment in children. They received (n=135; 15/group) root-canal treatment, pulpotomy, two- and one-surface restoration with and without local anesthesia; fluoride (with arch tray or cotton roll) or fissure sealant applications. Heart rate and SpO2 (peripheral oxygen saturation ) were monitored and The Facial Image Scale (FIS) and Children's Fear Survey Schedule-Dental subscales (CFSS-DS) were filled.

DETAILED DESCRIPTION:
The study was carried out following the approval by the local ethics committee (Malatya Clinical Studies Ethics Committee, 2017/76), and informed consent was signed by the parents. A total of 135 children (69 females 51.1%, 66 males 49.9%), aged 7-8 years (7.37±0.48 years), were admitted to Inonu University Faculty of Dentistry Department of Pediatric Dentistry. The study was planned with 135 children with 15 children in each group. For that purpose 9 groups were formed as 6 restorative and 3 protective applications. The restorative treatment groups included procedures with- and without-local anesthesia (LA). Procedures with LA included the groups as root canal treatment, pulpotomy, two-surface restoration and one-surface restoration. Procedures without LA included the groups as two-surface restoration and one-surface restoration. The protective application groups included the groups as fluoride application (by disposable arch tray or by cotton roll) and fissure sealant. The diagnosis and treatments were carried out by the same dentist (BA).Frankl's Behaviours Rating Scale (FBRS) is a method that is frequently used in studies based on the rating of behaviours. Children's attitudes during the dental examination were evaluated using FBRS. Behaviours of the child are examined in four groups in FBRS: definitely negative (Frankl-1), negative (Frankl-2), positive (Frankl-3), and definitely positive (Frankl-4).In terms of the standardization of the groups, only the children who were compatible with Frankl-3 or 4 classes were included in the study. Children with Farnkl-1 and -2 classes had negative compliance to treatment and therefore they were not included in the study. The patients were grouped according to treatment needs. Each patient who participated in the study was informed about the treatment to be applied to him/her and the measurements to be performed by using the tell-show-apply behavior method. Furthermore, the child informed the dentist about any discomforting stimuli by "raising his/her left hand up" and the dentist stopped when he/she received this warning. In the groups treated with local anesthesia, banana or strawberry flavored topical anesthetic gel (Vision Dental Pat Gel, WP Dental, Germany) that children might like was applied first. Then, the local anesthetic solution [Ultracain D-S ampoule (40 mg articain + 0.012 mg epinephrine) Aventis Pharma, Istanbul, Turkey] was injected by the traditional method with the help of a 2 cc set inject plastic dental injector (Tıbset Sterile Medical Equipment Industry Istanbul, Turkey). Only conventional root canal treatment and extirpation were planned for the children included in the root canal treatment group in the measurement session. In the groups to be treated with pulpotomy, it was noted that at least one of the approximal surfaces of the teeth had decay and iron sulfate (ViscoStat®, UltraDent, South Jordan, USA) was used as pulpotomy material. A Tofflemire matrix retainer and 0.05 mm thick matrix band (Hahnenkratt, Königsbach-Stein, Germany) were used in groups with a two-surface cavity. 2% NaF (Polimo® IMICRYL, Konya, Turkey) was preferred in groups who received fluoride application.

An aerator and micromotor were used as cavity preparation in the restorative treatment groups. Only the micromotor was used for polishing purposes in the protective treatment groups. FIS (Facial Image Scale) was assessed at three stages: at the moment they sat in the dental chair, 15 minutes after the start of the treatment, and 15 minutes after the end of the treatment. From the moment the patient sat in the dental chair, the probe of the bed-side monitor was attached to the patient's left index finger, and his/her heart rate and SpO2 (peripheral oxygen saturation ) of were monitored during the treatment period and the data were recorded. After the treatment of the patients was completed in that appointment, the CFSS-DS (Children's Fear Survey Schedule-Dental Subscales) was filled in by the patients under the supervision of their parents. In the mornings, 3 salivary samples were taken from the patients by their parents in the home environment, i.e. one day before the treatment, on the day of treatment and one day after the treatment. The non-stimulated total saliva was collected from the patients. The parents were warned about the fact that all of the three salivary samples should be taken at the 30th minute after awakening, between 07:00 and 07:30 am. Eating, drinking, brushing the teeth and using dental care products were not allowed. During the treatment period in the clinic, salivary samples were taken between 09.00 and 11.00 am. Saliva samples were taken in 3 stages, i.e. at the beginning of the treatment, at the 15th minute of the treatment, and 15 minutes after the end of the treatment. Sampling at 15th minute of the treatment process was standardized to correspond to the cavity with an aerator (at the enamel level) in restorative treatment groups and to the stage of polishing procedure with a micro motor in protective treatment groups. These measures were taken to prevent the saliva from contaminating the cavity.

ELIGIBILITY:
Inclusion Criteria:

* They were apparently healthy and had no previous experience of dental treatment
* In terms of the standardization of the groups, only the children who were compatible with Frankl-3 or 4 classes were included in the study.
* The patients were divided into groups taking into consideration the requirements of having no pain, abscess, fistula and no need for dental treatment requiring urgent intervention.

Exclusion Criteria:

* Patients, who did not meet the inclusion criteria for the study, who did not want to participate voluntarily, who ate and drank something 1 hour before the appointment, who used medication in the last 7 days, who used medication that may affect the salivary flow in the last 60 days or who left the dental treatment incomplete, were not included in the study.
* Children with Farnkl-1 and -2 classes had negative compliance to treatment and therefore they were not included in the study.

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Salivary cortisol levels at home | 30th minute after awakening, between 07:00 and 07:30 am.
  the day before treatment
Salivary cortisol levels at home | 30th minute after awakening, between 07:00 and 07:30 am.
  the treatment day
Salivary cortisol levels at home | 30th minute after awakening, between 07:00 and 07:30 am.
  the day after treatment
Salivary cortisol levels at clinic | beginning of the treatment, between 09:00 and 11:00 am.
  the treatment day
Salivary cortisol levels in clinic | 15th minute of the treatment, between 09:00 and 11:00 am.
  the treatment day
Salivary cortisol levels in clinic | 15th minute post treatment, between 09:00 and 11:00 am.
  the treatment day

CONTACTS AND LOCATIONS:
Overall Officials: Burçin Acar, Dr, Principal Investigator — Inonu University; Gulsum Duruk, Dr, Study Director — Inonu University; Sedat Yildiz, Prof., Study Chair — Inonu University; Cihat Uçar, Dr, Study Chair — Adiyaman University Research Hospital
Locations (1):
- Department of Pediatric Dentistry, Faculty of Dentistry, Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yfanti K, Kitraki E, Emmanouil D, Pandis N, Papagiannoulis L. Psychometric and biohormonal indices of dental anxiety in children. A prospective cohort study. Stress. 2014 Jul;17(4):296-304. doi: 10.3109/10253890.2014.918602. Epub 2014 May 27. PMID 24766350

DOCUMENTS (1):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT04338854/Prot_000.pdf